CLINICAL TRIAL: NCT05514184
Title: Plant-Focused Nutrition in Patients With Diabetes and Chronic Kidney Disease (PLAFOND Study): A Pilot/Feasibility Study
Brief Title: Plant-Focused Nutrition in Patients With Diabetes and Chronic Kidney Disease
Acronym: PLAFOND
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: VA Long Beach Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kamyar Kalantar-Zadeh, Professor of Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1750
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Disease (CKD) With Diabetes Mellitus (DM); CKD Stage 3; CKD Stage 4; CKD Stage 5; Diabetes Mellitus; Diabetic Kidney Disease
Keywords: plant-dominant low protein (PLADO) diet; plant-focused nutrition in CKD/DM (PLAFOND) diet; plant-based protein; glomerular hyperfiltration; high-protein diet; potassium restricted diet; renal disease progression; pilot/feasibility randomized controlled trial; diet adherence; meal plans; renal diet; Veterans; animal protein; continuous glucose monitoring (CGM); CKD-related symptoms; 24-hour urine nitrogen; Cystatin C and associated eGFR; dietary education; Medical Nutrition Therapy (MNT); uremic symptoms
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Diabetic Nephropathies | interventions — Diet

STUDY DESIGN:
Intervention Model Description: This is a pilot/feasibility, two-center (UCI and VA Long Beach), unblinded, randomized controlled trial, conducted in parallel with patients' routine CKD clinic visits, to test feasibility and safety of a patient-centered Plant-Focused Nutrition in CKD/DM (PLAFOND) comprised of >2/3 plant proteins compared to the standard-of-care renal diet, i.e., low K content with <1/3 plant protein.
Masking Description: Meal plans in both arms will be administrated by the study dietitians over 6-months among 120 patients with non-dialysis CKD/DM stages 3-5 for 6-months to examine dietary, nutritional, and glycemic endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-focused low-protein nutrition in diabetic CKD (PLAFOND) (Experimental): Participants randomized to this arm will receive PLAFOND dietary intervention consisting of a flexible low-protein meal plan including 0.6-0.8 g/kg/day dietary protein with >2/3% of the protein from plant-based sources, and the meal plan will be supported by dietitian who will provide dietary education and counseling to patients assigned to this arm.
  Interventions: Dietary Supplement: PLAFOND diet
- Standard-of-care renal diet (control group) (Active Comparator): Participants randomized to the control group will receive standard-of-care renal diet with low-potassium content based on dietitian counseling and guidance.
  Interventions: Dietary Supplement: PLAFOND diet

INTERVENTIONS:
Dietary Supplement: PLAFOND diet — PLAFOND is a pragmatic patient-centered dietary intervention supported by dietitians who provide education and counseling in the form of Medical Nutrition Therapy (MNT) consisting of 0.6-0.8 g/kg/day dietary protein with >2/3% of the protein from plant-proteins.
  Other Names: Plant-dominant low protein (PLADO) diet in the form of PLAFOND diet meal plans

SUMMARY:
In this pilot clinical trial, the investigators will recruit and randomize 120 patients with diabetes mellitus and chronic kidney disease (CKD/DM) stages 3 to 5 to a patient-centered and flexible Plant-Focused Nutrition in Diabetes (PLAFOND) diet with >2/3 plant-based sources, which will be compared with a standard-of-care CKD diet, which is usually a low-potassium and low-salt diet, over a 6-month period. Through this study, the investigators will determine whether the plant-focused diet intervention is feasible for patient adherence, whether this diet is safe by avoiding malnutrition, frailty, and high potassium or glucose blood levels, and whether patient reported outcomes are favorably impacted.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects 10-15% of US adults including 30-40% of persons with diabetes mellitus (DM), is associated with poor outcomes, and often progresses to requiring dialysis or transplantation. Half of all Americans with CKD also have DM. While traditional and emerging pharmacotherapies are often used in CKD with diabetes (CKD/DM), the synergistic role of dietary interventions has not been well examined. Low-carbohydrate low-fat diets are often recommended in DM, whereas low-protein diets (LPDs) are recommended for non-diabetic CKD with increasing emphasis on plant-based protein sources. Evidence suggests that high-protein diets with greater animal protein content may lead to glomerular hyperfiltration and faster decline in renal function in patients with CKD/DM. There remains major controversy regarding the potential risks vs. benefits of plant-based diets in CKD/DM, for which guidelines remain based on expert opinion. Given conventional dietary restrictions for the management of DM, there is concern that plant-based LPDs may lead to protein-energy wasting and hyperkalemia, whereas these diets may indeed be most beneficial in patients with CKD/DM given their faster rates of CKD progression as compared to non-diabetics. At present, clinical practice guidelines provide conflicting recommendations regarding the amount (low vs. high) and source (plant vs. animal) of dietary protein intake (DPI) in CKD/DM. Given that prior dietary trials in CKD such as the 1994 Modification of Diet in Renal Disease (MDRD) study excluded CKD/DM and did not examine the optimal proportion of plant vs. animal-based proteins, there is urgent unmet need for a rigorous dietary intervention study to examine the efficacy and safety of patient-centered plant-based diets in CKD/DM.

The investigators will conduct a pilot feasibility randomized controlled trial in parallel with patients' routine follow-up visits at ambulatory clinics to test the feasibility and safety of implementing a Plant- Focused Nutrition in CKD/DM (PLAFOND) diet with a DPI of 0.6-0.8 g/kg/d comprised of >2/3 plant-based sources, vs. standard-of-care renal diet with <1/3 plant-sources and low-potassium content, administrated by dietitians, over a 6-month period in 120 patients with CKD/DM stage 3-5. The investigators will determine whether the PLAFOND diet vs. the standard-of-care renal diet can be adhered to with consistent separation in dietary protein and plant-based proportions at 3- and 6-months. The investigators will also examine nutritional status, physical performance, and body composition, as well as glycemic measures using traditional metrics and continuous glucose monitoring, while other biochemical parameters and patient-reported outcomes including CKD-related symptoms will also be studied. In addition to providing the requisite feasibility and safety data of patient-conduct of future multi-center trials, this study will have major immediate impact by reinvigorating the critical role of dietary management of CKD/DM.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatient (>18 years old) with diabetes mellitus (DM), who attends ambulatory clinics in one of the two centers, who has the established diagnosis of stage 3-5 CKD and DM regardless of degree of proteinuria, and who wishes to prevent or delay dialysis initiation, is qualified, as long as there are at least 2 eGFRs <60 ml/min/1.73m2 three months apart with no intervening higher eGFR values.
* Participants will agree to follow the dietary instructions based on the randomization assignment and attend baseline visits as well as three additional ambulatory visits on Month 1, 3 and 6 post-randomization in person or via telehealth and respond to monthly or more frequent phone calls.

Exclusion Criteria:

* Having a terminal illness with a life expectancy <6 months such as stage 4 metastatic cancer.
* Patients with any serum potassium >5.5 mEq/L during the 6 months preceding the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Dietary adherence to PLAFOND vs. standard-of-care renal diet assessed by diet diaries | 6 months
  Dietary Adherence including separation in dietary plant-based proportions of >2/3 vs <1/3 at 3- and 6-months will be ascertained by 3-day diet diaries in all 120 participants as the primary outcome.

SECONDARY OUTCOMES:
Dietary adherence to PLAFOND vs. standard-of-care low-potassium renal diet assessed by 24-hour urine collections | 6 months
  Dietary Adherence and separation in dietary components of PLAFOND (plant-based proportions of protein >2/3) vs. low-potassium renal diet (<1/3 plant-based protein) at 3- and 6-months ascertained by and 24-hour urine collections (secondary outcome)
Physical function measured by Short Physical Performance Battery (SPPB) | 6 months
  Under "Nutritional and Physical Performance and Body Composition" physical function will be measured by Short Physical Performance Battery (SPPB), a value between 0 to 12 (higher suggesting more frail phenotype), at baseline, 3-, and 6-months.
Physical function measured by Fried Frailty Index | 6 months
  Under "Nutritional and Physical Performance and Body Composition" physical function will be measured by Fried Frailty Index, a score between 0 and 5, devided into ranking categories of non-frail (score 0), pre-frail (score 1-2) and frail (score 3-5), measured at baseline, 3-, and 6-months.
Muscle strength measured by handgrip strength | 6 months
  Under the "Nutritional and Physical Performance and Body Composition", muscle strength will be measured by handgrip strength using dynamometer, scored using force production in kilograms (0-90), at baseline, 3-, and 6-months.
Body composition using caliper anthropometry to measure mid-arm muscle circumference (MAMC) | 6 months
  Under "Nutritional and Physical Performance and Body Composition", body composition will be assessed using caliper anthropometry to measure mid-arm muscle circumference (MAMC) in cm (<12.5 cm as malnutrition), at baseline, 3-, and 6-months.
Body composition using near-infrared interactance | 6 months
  Under "Nutritional and Physical Performance and Body Composition", body composition will be assessed using caliper anthropometry and near-infrared interactance, producing percentage of body fat (unit: %), at baseline, 3-, and 6-months.
Biochemical parameter: serum A1c | 6 months
  Under "Glycemic, Renal and Safety Endpoints", biochemical parameter hemoglobin A1c, a value in percentage (normal rnage <5.5%), will be measured at baseline, and 1-, 3- and 6-months in all 120 participants
Biochemical parameter: serum potassium | 6 months
  Under "Glycemic, Renal and Safety Endpoints", biochemical parameter serum potassium, a valie in mEq/L (normal range: 3.5-5.3 mEq/L), will be measured at baseline, and 1-, 3- and 6-months in all 120 participants
Biochemical parameter: serum Cystatin C | 6 months
  Under "Glycemic, Renal and Safety Endpoints", biochemical parameter serum Cystatin C (mg/L) will be measured at baseline, and 1-, 3- and 6-months in all 120 participants
Biochemical parameter: urinary albumin to creatinine ratio (ACR) | 6 months
  Under "Glycemic, Renal and Safety Endpoints", biochemical parameters including hemoglobin A1c, potassium, and Cystatin C and albumin to creatinine ratio (ACR) in mg/g will be measured at baseline, and 1-, 3- and 6-months in all 120 participants
Glycemic status by continuous glucose monitoring (GCM) | 6 months
  Under "Glycemic Endpoints", glycemic status ascertained by continuous glucose monitoring (CGM) via DEXCOM will be examined in a substudy of 50 patients at baseline and at 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: Kamyar Kalantar-Zadeh, MD, MPH, PhD, Principal Investigator — University of California; Connie M Rhee, MD, MS, Principal Investigator — University of California
Locations (2):
- United States (2):
  - UCI, Orange, California
  - Harbor-UCLA/Lundquist, Torrance, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalantar-Zadeh K, Rhee CM, Joshi S, Brown-Tortorici A, Kramer HM. Medical nutrition therapy using plant-focused low-protein meal plans for management of chronic kidney disease in diabetes. Curr Opin Nephrol Hypertens. 2022 Jan 1;31(1):26-35. doi: 10.1097/MNH.0000000000000761. PMID 34750331
- [Background] Kalantar-Zadeh K, Joshi S, Schlueter R, Cooke J, Brown-Tortorici A, Donnelly M, Schulman S, Lau WL, Rhee CM, Streja E, Tantisattamo E, Ferrey AJ, Hanna R, Chen JLT, Malik S, Nguyen DV, Crowley ST, Kovesdy CP. Plant-Dominant Low-Protein Diet for Conservative Management of Chronic Kidney Disease. Nutrients. 2020 Jun 29;12(7):1931. doi: 10.3390/nu12071931. PMID 32610641
- [Background] Kalantar-Zadeh K, Fouque D. Nutritional Management of Chronic Kidney Disease. N Engl J Med. 2017 Nov 2;377(18):1765-1776. doi: 10.1056/NEJMra1700312. No abstract available. PMID 29091561
- [Background] Kalantar-Zadeh K, Jafar TH, Nitsch D, Neuen BL, Perkovic V. Chronic kidney disease. Lancet. 2021 Aug 28;398(10302):786-802. doi: 10.1016/S0140-6736(21)00519-5. Epub 2021 Jun 24. PMID 34175022
- [Background] Kistler BM, Moore LW, Benner D, Biruete A, Boaz M, Brunori G, Chen J, Drechsler C, Guebre-Egziabher F, Hensley MK, Iseki K, Kovesdy CP, Kuhlmann MK, Saxena A, Wee PT, Brown-Tortorici A, Garibotto G, Price SR, Yee-Moon Wang A, Kalantar-Zadeh K. The International Society of Renal Nutrition and Metabolism Commentary on the National Kidney Foundation and Academy of Nutrition and Dietetics KDOQI Clinical Practice Guideline for Nutrition in Chronic Kidney Disease. J Ren Nutr. 2021 Mar;31(2):116-120.e1. doi: 10.1053/j.jrn.2020.05.002. Epub 2020 Jul 29. PMID 32737016
- [Background] Kalantar-Zadeh K, Mattix-Kramer HJ, Moore LW. Culinary Medicine as a Core Component of the Medical Nutrition Therapy for Kidney Health and Disease. J Ren Nutr. 2021 Jan;31(1):1-4. doi: 10.1053/j.jrn.2020.11.002. No abstract available. PMID 33357519
- [Background] Rhee CM, Kalantar-Zadeh K, Moore LW. Medical Nutrition Therapy for Diabetic Kidney Disease. J Ren Nutr. 2021 May;31(3):229-232. doi: 10.1053/j.jrn.2021.03.004. No abstract available. PMID 33990265
- [Background] Kalantar-Zadeh K, Saville J, Moore LW. Unleashing the Power of Renal Nutrition in Value-Based Models of Kidney Care Choices: Leveraging Dietitians' Expertise and Medical Nutrition Therapy to Delay Dialysis Initiation. J Ren Nutr. 2022 Jul;32(4):367-370. doi: 10.1053/j.jrn.2022.05.001. Epub 2022 May 16. No abstract available. PMID 35589046